CLINICAL TRIAL: NCT00068809
Title: Short-Cycle Therapy in Adolescents Following Continuous Therapy With Established Viral Suppression: The Impact on Viral Load Suppression
Brief Title: 4-Day-A-Week Treatment Plan for HIV Infected Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATN 015 v 3.0
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: Treatment experienced; Treatment interruption
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Short-cycle therapy (SCT) (Experimental): At entry, subjects will switch from continuous HAART to SCT. All subjects will then be followed to assess viral load breakthrough over 48 weeks on SCT.
  Interventions: Procedure: Short Cycle Antiretroviral Therapy

INTERVENTIONS:
Procedure: Short Cycle Antiretroviral Therapy

SUMMARY:
This study will determine if taking anti-HIV drugs 4 days a week will control HIV-1 viral replication in patients who have already had at least 6 months of documented viral suppression with full-time treatment. If this strategy is shown to be safe in this study, a larger study will be undertaken to determine if the strategy can decrease overall drug exposure and help young people adjust more easily to a chronic medication schedule.

DETAILED DESCRIPTION:
HIV infected adolescents who require therapy face a lifetime of antiretroviral treatment. Highly active antiretroviral therapy (HAART) is associated with short- and long-term complications, and concerns are mounting about the cumulative effect of these complications as adolescents enter the third and fourth decade of life. A management strategy that can suppress the virus and decrease overall drug exposure is needed. In addition, the scheduling requirements for antiretroviral therapies interfere with the socialization and independence that an adolescent must accomplish to gain skills for a successful adult life. Not surprisingly, nonadherence to prescribed medications is common in teens. This multicenter, prospective, proof of concept trial will evaluate Short Cycle Therapy (SCT) in adolescents with sustained viral suppression of at least 6 months. While maintenance of viral load suppression can be viewed as either a safety or efficacy endpoint, the trial is constructed as an assessment of safety.

Eligible participants who have been on standard HAART therapy consisting of a Protease Inhibitor will switch to SCT therapy(4 days on treatment, 3 days off treatment each week) at entry. Participants will be seen in the clinic every other Monday during the first month, then monthly up to 24-weeks and then once every two months until the end of the 48-week study period. Plasma HIV RNA levels and CD4 cell counts will be performed at every visit. Medication adherence by self-report will be conducted every 2 weeks until week 24 and every 4-weeks thereafter until week 48. Fasting serum triglycerides and cholesterol will be measured at baseline, at week 24 and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Twelve to 24 years of age, regardless of the mode of transmission.
* Subjects must have been on a stable HAART regimen containing at least one PI and two NRTIs and no NNRTI for at least 3 months and be willing to continue the PI-containing regimen throughout the study period.
* Acceptable viral load defined as at least three plasma HIV-1 RNA levels ≤ 400 copies/ml within 12 months of study entry and no plasma HIV-1 RNA levels > 400 copies/ml within 6 months of entry date employing any clinically available viral load assay.
* Pre entry plasma HIV-1 RNA level <200 copies/ml by ultra-sensitive assay (Roche 1.5) within 30 days of study entry, performed in an assigned PACTG core virology laboratory.
* CD4+ T cell count >350 cells/microL within 30 days of study entry.
* Ability of subject and parent or legal guardian (when appropriate) to give written informed assent/consent and permission respectively.
* Subjects currently enrolled in ATN 015 Version 2.0 are eligible as follows:

  * Subjects randomized to standard continuous therapy (control arm). These subjects are eligible to be enrolled in ATN 015 Version 3.0 as new subjects if they meet the entry criteria for ATN Version 3.0. If eligible, they will be followed for the full 48 weeks.
  * Subjects randomized to short cycle therapy (experimental arm). These subjects are eligible to rollover to ATN 015 Version 3.0 and continue on SCT if they have not met a study endpoint. These subjects may not have a viral load value that meets a study endpoint (viz. a confirmed viral load of >400 copies/ml) and will continue on the intensive monitoring until they have completed 24 weeks when they will enter the less intensive 24 week phase of the study.
* Female subjects must be non-pregnant and willing to remain on effective contraception for the duration of the study. (Examples of acceptable forms of birth control include but are not limited to any form of hormonal contraception along with a barrier method, double barrier method, tubal ligation, or abstinence if it is the choice of the subject.)

Exclusion Criteria:

* On a HAART regimen containing an NNRTI or a HAART regimen with Abacavir (including Trizivir®).
* On any prohibited medication at the time of screening. Subjects with underlying reactive airway disease who are on either inhaled or brief, intermittent systemic steroids can be considered but their status must be reviewed with the protocol chair or vice chair through the standard ATN protocol query process.
* Active HIV-related opportunistic infection or any malignancy at the time of screening. (Female subjects who have been treated adequately for cervical dysplasia or CIN are eligible for study unless they are on systemic immunosuppressive therapy).
* Current treatment for known or suspected active serious bacterial infection.
* Pregnancy.
* Any laboratory abnormalities Grade 3 or greater as defined in Appendix III at the time of screening.
* Subjects receiving pharmacological treatment for elevated cholesterol and triglyceride levels.

If a candidate fails the eligibility criteria (inclusion or exclusion), she or he may be screened again for eligibility after a period of 30 days.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2003-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Assess VL Suppression for Subjects on SCT over a 24 Week and 48 Week Period | 48 Weeks
  To assess viral load suppression (≤ 400 copies/ml) for subjects on SCT over a 24 week and a 48 week period.
  The primary endpoint is defined as the time of confirmed VL > 400 copies/ml at any time after study entry up to and including the 48th week of follow-up.

SECONDARY OUTCOMES:
Assess CD4+ T-cell count over time for subjects on SCT from baseline to week 48 | 48 Weeks
  To assess CD4+ T-cell count over time for subjects on SCT from baseline to week 48. These values will be compared at (1) the period of time from study entry to viral load rebound (> 400 copies/ml), (2) the period of time from study entry to subject dropout, or (3) the period of time from study entry to administrative end of study at 48 weeks, depending on each subject's disposition.
Compare differences in various values from study entry to Weeks 24 and 48 | 48 Weeks
  To compare differences in fasting cholesterol, triglycerides, LDL, HDL, and VLDL levels from study entry to weeks 24 and 48
Assess the adherence level over time | Week 48
  To assess the adherence level over time using the PACTG Pediatric Adherence Questionnaire Module I, every two weeks up to week 24 and every four weeks until week 48
Assess genotypic resistance as necessary | 48 Weeks
  To assess subject-specific plasma genotypic resistance for subjects with viral load >1000 copies/ml at time of viral load rebound.

CONTACTS AND LOCATIONS:
Overall Officials: Bret J Rudy, MD, Study Chair — Children's Hospital of Philadelphia, The University of Pennsylvania School of Medicine
Locations (9):
- United States (8):
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - Stoger Hospital of Cook County, Chicago, Illinois
  - Mt. Sinai Hospital, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- See also: Description of Adolescent Trials Networks (ATN) and contact information — http://www.atnonline.org